CLINICAL TRIAL: NCT05342090
Title: Randomized Controlled Trial of Standardized Counselling on Postoperative Return to Sexual Activity After Pelvic Reconstructive Surgery
Brief Title: Postoperative Return to Sexual Activity
Acronym: PoRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Wisconsin, Madison (Other); Albany Medical College (Other); Penn State University (Other); Columbia University (Other); University of Chicago (Other); University of Florida (Other); WellSpan Health (Other); University of New Mexico (Other); Weill Medical College of Cornell University (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Shunaha Kim-Fine, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-0749
Record Dates: First submitted 2022-03-30; First posted 2022-04-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Sexual Function Disturbances; Pelvic Organ Prolapse; Stress Urinary Incontinence; Surgery
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized Counselling Tool (Active Comparator): If randomized to the treatment group, patients will be counselled using the structured counselling tool, and given a bulleted list of the counseling instrument to take home with them.
  Interventions: Other: Structured Counselling Tool
- Control (No Intervention): Routine postoperative counselling and care will be administered with no specific standardized counselling for return to sexual activity after surgery.

INTERVENTIONS:
Other: Structured Counselling Tool — Participants will be administered a Structured Counselling Tool that addresses the following themes: outside influences, conflicting emotions, uncertainty, sexual changes and stability, normalization, self-image
  Arms: Standardized Counselling Tool

SUMMARY:
To determine if standardized counselling regarding first sexual encounter after pelvic reconstructive surgery for pelvic organ prolapse and / or urinary incontinence improves postoperative preparedness to return to sexual activity and sexual function.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial comparing standardized counselling to routine counseling regarding return to sexual activity using a previously developed structured counselling instrument. Adult women (age ≥18 years) who are undergoing reconstructive surgery for pelvic organ prolapse and / or urinary incontinence who report that they are currently sexually active (as defined by their own assessment of the meaning of this question) will be eligible to participate and recruited during their preoperative visit. The recruitment will take place across 10 sites in Canada and the Unites States. The hypothesis is that use of a newly developed standardized counselling intervention regarding resumption of sexual activity will result in improved preparedness to return to sexual function compared to routine care. The primary outcome will be preparedness at 2-6 months postoperatively. Preparedness for return to sexual activity will be measured by modifying the Patient Preparedness Questionnaire, Question #11: "Overall, I feel prepared for my upcoming surgery" to make it relevant to sexual activity following surgery. The investigators will consider women prepared if they answer "strongly agree" on a 6-point Likert scale from "strongly agree" to "strongly disagree" to the modified statement: "Overall, I feel prepared for resuming sexual activity after my surgery". In addition to the primary outcome, the investigators will compare the secondary outcomes of sexual function, time to return to sexual activity, and postoperative pain with sexual activity. Sexual function will be measured by Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) score. Pain with sexual activity will be assessed by response to question 11 on PISQ-IR: "How often do you feel pain during sexual intercourse?" Women who have already consented for surgery for pelvic organ prolapse surgery will be approached to offer participation in the study at the pre-operative visit. After enrollment in the study, women will complete demographic information, undergo a pelvic organ prolapse quantification examination, and complete the PISQ IR and the Pelvic Floor Distress Inventory - 20 (PFDI-20).

Women will then be randomized to either usual or scripted counseling for resumption of sexual activity. The randomization assignment will occur as close to the intervention as possible, i.e. the night before, or the morning of, scheduled 6-8 week postoperative appointment. The randomization schema will be generated using an online randomization table with alternating blocks of 4 and 6. If randomized to the treatment group, patients will be counselled using the structured counselling instrument, and given a bulleted list of the counseling instrument to take home with them. After the visit, women will complete the PFDI-20 and Preparedness question in telephone-administered, paper or online questionnaire format.

The study team will contact each participant by telephone or electronically at 1 month intervals starting at 2 months after surgery, to ascertain whether they had returned to sexual activity. If the postoperative visit occurred at 8 weeks, the first contact will occur at 3 months. If the patient has returned to sexual activity, again defined by the patient's own interpretation of the question about return to sexual activity, then women will be asked to complete the PISQ-IR and Preparedness question by telephone-administered, mailed paper, or online questionnaire format. No further followup will be required after return to sexual activity. If women are not yet returned to sexual activity, they will be contacted at 1 month intervals, to a maximum interval of 6 months after surgery, to determine return to sexual activity and timing of administration of the PISQ-IR and Preparedness question. If a woman has not yet returned to sexual activity by 6 months, we will administer the PISQ-IR and Preparedness question by telephone-administered, mailed paper, or online questionnaire format.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (age ≥ 18 years)
* consented for pelvic reconstructive surgery for pelvic organ prolapse and / or urinary incontinence
* currently sexually active as defined by self-report
* able to speak and read English

Exclusion Criteria:

* Not currently sexually active as defined by self-report
* vulvar dermatologic pathology (Lichen sclerosus, lichen planus)
* chronic pelvic pain
* unable to consent or complete outcomes due to mental incapacity, prisoners or incarcerated women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Preparedness to return to sexual activity | 2-6 months postoperative
  Preparedness for return to sexual activity will be measured by modifying the Patient Preparedness Questionnaire, Question #11: "Overall, I feel prepared for my upcoming surgery" to make it relevant to sexual activity following surgery. We will consider women prepared if they answer "strongly agree" on a 6-point Likert scale. The scale ranges from "strongly agree" to "strongly disagree" to the modified statement: "Overall, I feel prepared for resuming sexual activity after my surgery".

SECONDARY OUTCOMES:
Sexual Function | 2-6 months postoperative
  Sexual function will be measured by Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) score. Higher scores indicate better sexual function.
  Scores can range from 0 to 125. Pain with sexual activity will be assessed by response to question 11 on PISQ-IR: "How often do you feel pain during sexual intercourse?" Possible responses to this question are: "Never", "Rarely", "Sometimes", "Usually", "Always"
Postoperative Pain | 2-6 months postoperative
  Postoperative pain will be evaluated with responses to the question: "Have you experienced pain in your pelvis in the last week (7 days)?" Responses of "yes" and "no" will be recorded
Time to Return to Sexual Function | 2-6 months postoperative
  Time to Return to Sexual Function will be determined by responses to self-report of date of return to sexual activity after surgery. The duration of time between surgery and return to sexual activity will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Shunaha Kim-Fine, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Health Services, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No identifiers will be shared among co-investigators or other researchers. This is because the information is stored in Redcap and site PIs and their research staff will only have access to IPDs in their own institution but not across outside institutions.

REFERENCES:
- [Background] Samuelsson EC, Victor FT, Tibblin G, Svardsudd KF. Signs of genital prolapse in a Swedish population of women 20 to 59 years of age and possible related factors. Am J Obstet Gynecol. 1999 Feb;180(2 Pt 1):299-305. doi: 10.1016/s0002-9378(99)70203-6. PMID 9988790
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Dunivan GC, McGuire BL, Rishel Brakey HA, Komesu YM, Rogers RG, Sussman AL. A longitudinal qualitative evaluation of patient perspectives of adverse events after pelvic reconstructive surgery. Int Urogynecol J. 2019 Dec;30(12):2023-2028. doi: 10.1007/s00192-019-03998-7. Epub 2019 Jun 11. PMID 31187179
- [Background] Antosh DD, Kim-Fine S, Meriwether KV, Kanter G, Dieter AA, Mamik MM, Good M, Singh R, Alas A, Foda MA, Balk EM, Rahn DD, Rogers RG. Changes in Sexual Activity and Function After Pelvic Organ Prolapse Surgery: A Systematic Review. Obstet Gynecol. 2020 Nov;136(5):922-931. doi: 10.1097/AOG.0000000000004125. PMID 33030874
- [Background] Kenton K, Pham T, Mueller E, Brubaker L. Patient preparedness: an important predictor of surgical outcome. Am J Obstet Gynecol. 2007 Dec;197(6):654.e1-6. doi: 10.1016/j.ajog.2007.08.059. PMID 18060968
- [Derived] Kim-Fine S, Caldwell L, Long J, Meriwether KV, Iyer S, Heisler CA, Hudson P, Husk K, Lozo S, Demtchouk V, Huang B, Antosh DD, Rogers RG; Society of Gynecologic Surgeons Consortium of Research in Pelvic Surgery. Intervention Counseling for Return to Sex After Urogynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2025 Nov 1;146(5):701-709. doi: 10.1097/AOG.0000000000006064. Epub 2025 Sep 11. PMID 40934518
- [Derived] Caldwell L, Kim-Fine S, Antosh DD, Husk K, Meriwether KV, Long JB, Heisler CA, Hudson PL, Lozo S, Iyer S, Weber LeBrun EE, Rogers RG. Standardized Counseling Tool for Returning to Sexual Activity After Pelvic Reconstructive Surgery. Obstet Gynecol. 2025 Nov 1;146(5):e80-e84. doi: 10.1097/AOG.0000000000005938. Epub 2025 Jun 13. PMID 40505118